CLINICAL TRIAL: NCT02459340
Title: Effectiveness of Therapeutic Treatment: Hot and Cold Self-regulation in Posttraumatic Stress Disorder and Dissociative Disorder
Brief Title: Emotional and Cognitive Self-regulation, an EEG Study
Acronym: ECSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yolanda Schlumpf, PhD (Other)
Collaborators: Clienia Littenheid AG (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Yolanda Schlumpf, PhD, PhD, Clienia Littenheid AG
Organization: Clienia Littenheid AG (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLUZH-1
Record Dates: First submitted 2015-05-11; First posted 2015-06-02 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Complex Posttraumatic Stress Disorder (cPTSD); Dissociative Disorder Not Otherwise Specified (DDNOS); Dissociative Identity Disorder (DID)
MeSH Terms: conditions — Dissociative Identity Disorder | interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient group (Experimental): Inpatient setting (cPTSD, DDNOS, DIS): Trauma-adapted psychotherapy (individual and group setting), body-related, cognitive stabilization groups, pharmacotherapy, and other non-verbal treatment modalities (e.g. music, art, and occupational therapy)
  Interventions: Other: therapeutic treatment (inpatient and outpatient setting)
- healthy control group (No Intervention): passive control group

INTERVENTIONS:
Other: therapeutic treatment (inpatient and outpatient setting)
  Arms: patient group

SUMMARY:
The main goal of the proposed project is to assess treatment-induced changes of electrophysiological and psychophysiological correlates of the capacity to regulate emotion, executive functions, and clinical measures in individuals with complex posttraumatic stress disorder and dissociative disorders in a naturalistic inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

-ability to undergo EEG measurement/psychophysiological measurement

Exclusion Criteria:

* regular substance use
* acute suicidality
* comorbid psychosis

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
event-related potential (ERP) | up to 6 months
power in specific frequency bands | up to 6 month

SECONDARY OUTCOMES:
heart rate | up to 6 months
electrodermal activity | up to 6 months
executive function | up to 6 months
  working memory, Schuhfried test battery
measurement of psychological symptoms | up to 6 month
  questionnaire, Brief Symptom Inventory (BSI)
assessment of emotion regulation and dysregulation | up to 6 month
  questionnaire, Difficulties in Emotion Regulation Scale (DERS)

CONTACTS AND LOCATIONS:
Overall Officials: Silke Bachmann, Prof. Dr. med., Study Director — Privat Clinic Clienia Littenheid; Yolanda Schlumpf, PhD, Principal Investigator — Privat Clinic Clienia Littenheid, University of Zurich
Locations (1):
- Privat Clinic Clienia Littenheid, Littenheid, Thurgau, Switzerland

REFERENCES:
- [Derived] Schlumpf YR, Nijenhuis ERS, Klein C, Jancke L, Bachmann S. Functional connectivity changes in the delta frequency band following trauma treatment in complex trauma and dissociative disorder patients. Front Psychiatry. 2022 Jul 25;13:889560. doi: 10.3389/fpsyt.2022.889560. eCollection 2022. PMID 35966482
- [Derived] Schlumpf YR, Nijenhuis ERS, Klein C, Jancke L, Bachmann S. Resting-state functional connectivity in patients with a complex PTSD or complex dissociative disorder before and after inpatient trauma treatment. Brain Behav. 2021 Jul;11(7):e02200. doi: 10.1002/brb3.2200. Epub 2021 Jun 9. PMID 34105902